CLINICAL TRIAL: NCT02405013
Title: TAC (Treatment Africa Hepatitis C) : Feasibility, Tolerance and Efficacy of Interferon-free, Antiviral Treatment With Sofosbuvir + Ribavirin for the Treatment of Genotype 2 and Sofosbuvir/Ledipasvir for the Treatment of Genotype 1 and 4 Hepatitis C Virus-infected Patients in West and Central Africa
Brief Title: Feasibility, Tolerance and Efficacy of Interferon-free, Antiviral Treatment With Sofosbuvir + Ribavirin for the Treatment of Genotype 2 and Sofosbuvir/Ledipasvir for the Treatment of Genotype 1 and 4 Hepatitis C Virus-infected Patients in West and Central Africa
Acronym: TAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12311 TAC
Record Dates: First submitted 2015-02-20; First posted 2015-04-01 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C; HIV Infection
Keywords: Africa; Hepatitis C; HIV; Antiviral treatment; Adults; HCV genotype 1; HCV genotype 2; HCV genotype 4
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — Sofosbuvir; Ribavirin; ledipasvir, sofosbuvir drug combination; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sofosbuvir+Ribavirin (Experimental): Sofosbuvir 400mg QD (Sovaldi®) + Ribavirin weight-adjusted dosing (1000mg BID in patients < 75kg and 1200mg BID in patients ≥ 75kg) in treatment-naïve patients infected with HCV genotype 2 (12-week course)
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin
- Sofosbuvir+Ledipasvir (Experimental): Sofosbuvir/Ledipasvir 400mg/90mg (Harvoni®) in treatment-naïve patients infected with HCV genotype 1 or genotype 4 (12-week course)
  Interventions: Drug: Sofosbuvir; Drug: Ledipasvir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400mg QD (Sovaldi®) in treatment-naïve patients infected with HCV genotype 2 (12-week course)
  Other Names: Sovaldi®
  Arms: Sofosbuvir+Ribavirin
Drug: Ribavirin — Ribavirin weight-adjusted dosing (1000mg BID in patients < 75kg and 1200mg BID in patients ≥ 75kg) in treatment-naïve patients infected with HCV genotype 2 (12-week course)
  Arms: Sofosbuvir+Ribavirin
Drug: Sofosbuvir — Sofosbuvir/Ledipasvir 400mg/90mg (Harvoni®) in treatment-naïve patients infected with HCV genotype 1 or genotype 4 (12-week course)
  Other Names: Harvoni®
  Arms: Sofosbuvir+Ledipasvir
Drug: Ledipasvir — Sofosbuvir/Ledipasvir 400mg/90mg (Harvoni®) in treatment-naïve patients infected with HCV genotype 1 or genotype 4 (12-week course)
  Other Names: Harvoni®
  Arms: Sofosbuvir+Ledipasvir

SUMMARY:
Primary Objective:

To evaluate the efficacy (sustained virological response 12 weeks after end-of-treatment [SVR12]) of 12-week course of an interferon-free regimen combining sofosbuvir and weight-dosed ribavirin (genotype 2), or sofosbuvir and ledipasvir (genotype 1 or 4) in treatment-naïve patients infected with HCV genotype 1, 2 or 4 in West and Central Africa

Secondary Objectives:

1. To estimate the study treatment SVR24 rate
2. To evaluate the clinical and biological tolerance of study treatment
3. To describe HCV kinetics under HCV treatment, and identify associated factors
4. To describe the evolution of HIV disease under HCV treatment in HVC-HIV co-infected patients
5. To describe the changes of liver fibrosis based on non-invasive tests between treatment initiation, week 24, and week 36 after treatment, and estimate its association with SVR12 or SVR24
6. To identify factors associated with SVR12 and SVR24 (including HIV status)
7. To evaluate the performance of a nanodevice for rapid diagnosis of HCV viral load and genotypying and for assessing response to treatment (SVR12 and SVR24)
8. Facilitate the detection and treatment of those infected with HCV by supporting national initiatives for access to strategies without interferon
9. To set up a HCV clinical research network across French and English-speaking African countries, able to run large-scale comparative randomized clinical trials in a near future.

DETAILED DESCRIPTION:
Study design Multicenter, phase IIb, non randomized, open-label trial involving 3 groups of HCV-mono infected or HCV-HIV co-infected patients: group G1 (patients infected with HCV genotype 1), group G2 (patients infected with HCV genotype 2), and group G4 (patients infected with HCV genotype 4).

Number of Subjects A sample size of 40 patients per group will allow to demonstrate that the SVR12 is >70% ("expected efficacy" in difficult-to-treat patients, according to SPARE interim results), with the lower bound of the confidence interval being >50% ("unacceptable" efficacy). The overall sample size is 3x40=120 patients.

Participating Countries 3 countries from West Africa (Senegal, Côte d'Ivoire) and Central Africa (Cameroon) Number of Sites 5 clinical sites:

* Côte d'Ivoire: Hepatology Departementat the Yopougon University Teaching Hospital, , Abidjan; and Blood Donors clinic (CMSDS) at the National Blood Bank (CNTS), Abidjan
* Senegal: CRCF (Centre Régional de Recherche et de Formation), and Fann University Teaching Hospital
* Cameroon: Clinique de la Cathédrale

Duration of Recruitment : 6 months

Duration of Treatment : 12 weeks

Duration of follow-up : 36 weeks

Anticipated Start Date / Anticipated End Date: November 2015 - October 2016

Target Population /Demographics : Patients >18 years, living with chronic hepatitis C genotype 1, 2 or 4, in West and Central Africa. In each genotype group approx. 50% of patients will be HCV-HIV co-infected, and 50% of patients will be mono-infected with HCV

This study will enable us to assess the feasibility, tolerance and efficacy of such a strategy in resource-constrained settings with considerable treatment needs.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Confirmed G1, G2 or G4 HCV infection
* Plasma HCV-RNA ≥1000 IU/mL
* No history of HCV treatment of any kind
* Willingness to use a birth control method (hormonal or intrauterine device for women, condoms for men), starting before HCV treatment initiation and continued until 4months (women) and 7 months (men) after end of treatment.
* Weight ≥40 kg and ≤125 kg

For patients infected with HIV :

* Confirmed HIV-1 infection
* Stable HIV treatment for at least 8 weeks with two NRTIs (tenofovir or abacavir, and lamivudine or emtricitabine) and a third agent (raltegravir, lopinavir/ritonavir, atazanavir/ritonavir, darunavir/ritonavir, efavirenz, nevirapine)
* Current CD4+ lymphocytes count ≥100/mm3
* Current plasma HIV-1 RNA <200 copies/mL

Exclusion Criteria:

For each patient:

* Cirrhosis classified Child-Pugh B or C
* Co-infection by the Hepatitis B virus
* Pregnant or breastfeeding ongoing
* History of transplantation of organs or tissues
* Progressive Cancer, including hepatocellular carcinoma
* Epilepsy
* Sickle Cell Disease
* A history of myocardial infarction or other severe heart disease
* Excessive consumption of alcohol or drug users, in the absence of substitution by methadone, a stable weaning for more than three months should be required
* Ongoing Participation in another clinical trial
* Contraindications to the Sofosbuvir as defined in the Summary of Product Characteristics
* At least one of the following laboratory abnormalities:

Haemoglobin <10 g / 100 ml (woman) <11 g / 100 ml (man) Platelet count <50,000 / mm3 polymorphonuclear neutrophils rate <750 / mm3 Creatinine clearance <50ml / min

For patients infected with HIV:

* Severe opportunistic infections in the last 6 months
* Poor adherence to antiretroviral treatment history
* Use of antiretroviral drugs other than those permitted in the test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Load Response (SVR) | Week 12

SECONDARY OUTCOMES:
Tolerance | 36 weeks
  Grade 1, 2, 3 and 4 clinical or biological events (ACTG grading table), Adverse events-related HCV treatment discontinuation Adverse events-related ARV treatment modification
Viral kinetics as measured by SVR 24 and HCV-RNA | W0, W2, W4, W12, W24, W36
  SVR 24 and HCV-RNA
HIV treatment clinical parameters | 36 weeks
  Number, nature and incidence of severe morbid events related to HIV, and clinical and biological events of grade 3 or 4 (ANRS scale) related to the ARV treatment
Liver fibrosis | W0, W24 and W36
  Elastometry score and only for cirrhotic patients : Child-Pugh score
Adherence measured by number of remaining tablets at each visit based on the number of tablets should have been taken as a percentage of the total dose | W4, W8, W12
  Number of remaining tablets at each visit based on the number of tablets should have been taken as a percentage of the total dose
Quality of life | 36 weeks
  proportion of people reporting symptoms in the scale of symptoms experienced (scale of side effects perception SF12)
Performance of an unit of nanotechnology | 36 weeks
  calculation of sensitivity / specificity / positive predictive value and negative of each of the steps that will be performed (genotype, viral load) compared to the reference measurement (PCR for viral load and sequencing to genotype).
Setting up the network: | 36 weeks
  number of network meetings that have taken place before the end of the trial, the number of training sessions (on site or online) and the numbers enrolled in the network active partners. The ultimate goal is the establishment of an e-learning platform that will be an ancillary project.
Integration Access initiatives evaluated by the number of patients off protocol that will have access to new anti-HCV treatment due to "ACCESS" programs of pharmaceutical companies conducting such programs in Sub-Saharan Africa | 36 weeks
  It will be evaluated by the number of patients off protocol that will have access to new anti-HCV treatment due to "ACCESS" programs of pharmaceutical companies conducting such programs in Sub-Saharan Africa
Biological events | W0, W24 and W36
  Plasma HIV-RNA and CD4 count

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Moh, Dr, Study Director — Programme PACCI; Babacar Sylla, Study Director — Institut de Médecine et d'Epidémiologie Appliquée
Locations (4):
- Clinique de la Cathédrale, Yaoundé, Cameroon
- Côte d’Ivoire (2):
  - Centre de suivi des donneurs de sang, Abidjan
  - CHU de Youpougon - Service de Gastro-entéro-hépatologie, Abidjan
- CHU Fann, Service des Maladies Infectieuses, Dakar, Senegal

REFERENCES:
- [Derived] Marcellin F, Mourad A, Lemoine M, Kouanfack C, Seydi M, Carrieri P, Attia A, Protopopescu C, Lacombe K, Boyer S. Patient-reported outcomes with direct-acting antiviral treatment for hepatitis C in West and Central Africa (TAC ANRS 12311 trial). JHEP Rep. 2022 Dec 28;5(3):100665. doi: 10.1016/j.jhepr.2022.100665. eCollection 2023 Mar. PMID 36686592